CLINICAL TRIAL: NCT03937037
Title: Effect of Intermittent Saline Irrigation in Reducing Choledocholithiasis Recurrence After ERCP
Brief Title: Effect of Saline Irrigation in Reducing Choledocholithiasis Recurrence After ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, M.D., Ph. D, Direct of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Saline irrigation follow-up
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Stone - Biliary
Keywords: ERCP; Common bile duct stone; Cholangitis; Residual stone; Irrigation; Recurrence
MeSH Terms: conditions — Cholecystolithiasis; Gallstones; Cholangitis; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline irrigation (Experimental): CBD stone removal after routine ERCP procedure,100ml saline irrigation after a balloon occlusion cholangiogram confirming the absence of stones.
  Interventions: Procedure: Saline irrigation
- None saline irrigation (No Intervention): CBD stone removal after routine ERCP procedure, a balloon occlusion cholangiogram confirms the absence of stones.

INTERVENTIONS:
Procedure: Saline irrigation — 100ml saline irrigation after CBD stone removal with routine ERCP procedure
  Arms: Saline irrigation

SUMMARY:
In this prospective study, the investigators assessed the utility of intermittent saline irrigation in reducing the recurrent rate of choledocholithiasis after the endoscopic extraction for common bile duct stones, and it does not increase the rate of procedure-related complications.

DETAILED DESCRIPTION:
In recent years, an endoscopic retrograde cholangiopancreatography (ERCP) is the golden standard procedure to remove the common bile duct stones(CBD). Nevertheless, it is reported that the recurrence rate of CBD stones is 4% to 24% after ERCP. The contributing factors were periampullar diverticulum, situ gallbladder, and incomplete CBD stone clearance. The main reason of stone recurrence is incomplete CBD stone clearance including remnant stone fragments themselves and tinny fragments can act as a nidus for further CBD stone growth. It is difficult to retrieve these fine fragments completely using conventional devices such as retrieval basket and ballon. Therefore, the investigators attempt to remove residual stone fragments by means of saline infusion. Saline irrigation has many advantages such as better effect and less side effect and no extra cost. It is reported that use intraductal ultrasonography (IDUS) to demonstrate residual CBD stones. However, IDUS has limited availability in clinical practice. The single-operator cholangioscopy (SOC)-system gains widespread acceptance because of its independent washing channels and direct viewing.

The purpose of this study is to evaluate whether saline solution irrigation would decrease the recurrent rate of choledocholithiasis after endoscopy retrieval stones.

ELIGIBILITY:
Inclusion Criteria:

* With ERCP indications
* With mechanical lithotripsy during operation

Exclusion Criteria:

* Unwillingness or inability to consent for the study
* Unstable vital signs
* Coagulation dysfunction (INR>1.5) and low peripheral blood platelet count (<50×10 ^9 / L) or using anti-coagulation drugs
* Prior surgery of Bismuth Ⅱ, Roux-en-Y and cholangiojejunostomy
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease (such as decompensated liver cirrhosis, liver failure and so on), septic shock
* Biliary-duodenal fistula confirmed during ERCP
* Pregnant women or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Recurrence of CBD Stones | 3 years
  Number of Participants with stones detected by Magnetic resonance cholangiopancreatography, CT or US confirms CBD stone recurrence no matter symptomatic choledocholithiasis or not

SECONDARY OUTCOMES:
Number of Participants with Cholangitis | 3 years
  Temperature should be more than 38 ℃, with right upper abdominal pain, blood routine showing the total amount of the White Blood Cell (WBC), and the amount of polymorphonuclear neutrophil(PMN) are above normal
Number of Participants with Pancreatitis | 3 years
  Typical abdominal pain, with the level of serum amylase increasing at least 3 times of the normal range within 24 hours after surgery, and there are also radiographic evidence suggesting the shape of pancreas has changed
Number of Participants with Bleeding | 1 month
  Was defined as the clinical and endoscopic evidence of hemorrhage associated. with a decreasing the hemoglobin level >2 g/dl
Number of Participants with Perforation | 1 month
  Was defined as the presence of air or contrast in the retroperitoneal space
Procedure time of each case | 7 days
  From the moment the endoscope entered, to the moment withdraw the scope

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, MD,PhD, Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn DW, Lee SH, Paik WH, Song BJ, Park JM, Kim J, Jeong JB, Hwang JH, Ryu JK, Kim YT. Effects of Saline Irrigation of the Bile Duct to Reduce the Rate of Residual Common Bile Duct Stones: A Multicenter, Prospective, Randomized Study. Am J Gastroenterol. 2018 Apr;113(4):548-555. doi: 10.1038/ajg.2018.21. Epub 2018 Mar 27. PMID 29610513
- [Background] Ang TL, Teo EK, Fock KM, Lyn Tan JY. Are there roles for intraductal US and saline solution irrigation in ensuring complete clearance of common bile duct stones? Gastrointest Endosc. 2009 Jun;69(7):1276-81. doi: 10.1016/j.gie.2008.10.018. Epub 2009 Feb 26. PMID 19249039
- [Derived] Lin Y, Yang M, Cao J, Zhang X, Mi N, Yang X, Wang H, Gao L, Bai M, Fu W, Li X, Yue P, Yuan J, Meng W, Leung JW. Saline irrigation for reducing the recurrence of common bile duct stones after lithotripsy: a randomized controlled trial. EClinicalMedicine. 2023 Apr 27;59:101978. doi: 10.1016/j.eclinm.2023.101978. eCollection 2023 May. PMID 37152367